CLINICAL TRIAL: NCT02859220
Title: Study of the Influence of Dosages of 1-84 and 7-84 Fragments of PTH Compared to Conventional Dosage on the Balance of Calcium and Phosphate in Hemodialysis
Brief Title: Study of the Influence of Dosages of 1-84 and 7-84 Fragments of Parathyroid Hormone Compared to Conventional Dosage on the Balance of Calcium and Phosphate in Hemodialysis (PTH)
Acronym: PTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: BRD/05/12-C
Record Dates: First submitted 2011-06-29; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2011-06

CONDITIONS: Hemodialysis Patients
Keywords: hemodialysis; PTH

ARMS (2):
- group 1 (Other): group 1 : Roche Elecsys intact PTH
  Interventions: Other: Determination of PTH following
- group 2 (Other): group 2 : PTH 1-84 complete (PAC) report and CAP / PTH 7-84 (CIP), Duo PTH IRMA Scantibodies
  Interventions: Other: Determination of PTH following:

INTERVENTIONS:
Other: Determination of PTH following — Determination of PTH following:
  in group 1: intact PTH Elecsys Roche
  Arms: group 1
Other: Determination of PTH following: — PTH 1-84 complete (PAC) report and CAP / CIP, the package "Duo PTH IRMA Scantibodies." The CIP is obtained by calculating the difference between total intact PTH and PTH 1-84 in the kit used.
  Arms: group 2

SUMMARY:
This study included 80 patients with end stage renal disease requiring dialysis treatment to evaluate two techniques for the determination of parathyroid hormone (PTH)

Objective: To evaluate whether the monitoring of hemodialysis patients by measurement of PTH 1-84 Complete (CAP =cyclase activating PTH) and the ratio (1-84 PTH (CAP)/7-84 PTH (CIP = cyclase inactivating PTH) with kit "Duo PTH Immunoradiometric Scantibodies" allows an improvement in the therapeutic management of abnormal calcium and phosphate, with a better match to the targets of current international recommendations, followed by the conventional intact PTH assay.

Primary endpoint:

For each patient, a score will be awarded based on the number of criteria (including calcium, phosphorus and calcium phosphate product) in the target international guidelines :0-1-2 or 3.

The primary endpoint will be the average scores in both groups at the beginning and the end of the study,

Main secondary endpoints:

* Changes in the number of patients responding to international guidelines for each of the three parameters studied (serum phosphate, corrected calcium, phosphorus product) in the 2 groups,
* Evolution of Elecsys intact PTH Roche in the 2 groups,
* Salaries and changes in the number of drugs to normalize the phospho-calcium balance in each group received,
* cardiovascular events (morbidity and cardiovascular mortality),
* Total mortality.

Statistical analysis:

This is a randomized, two parallel arms. The investigators will compare the average number of criteria on calcium and phosphate in the target according to a Mann-Whitney. The analysis will be performed with the software Splus.

ELIGIBILITY:
Inclusion Criteria:

* replacement therapy by hemodialysis for at least three months in the hemodialysis center of Nantes University Hospital,
* intact PTH ≥ 100 pg / mL during the visit of inclusion.

Exclusion Criteria:

* intact PTH <100 pg / mL during the visit of inclusion
* Life expectancy estimated at less than one year at the time of inclusion, because of a disease diagnosed prior to the initiation of the study,
* bone pathology diagnosed prior to the initiation of the study that interfere with calcium and phosphate metabolism (myeloma, Paget ...).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
improving the therapeutic management of calcium and phosphate abnormalities by conventional PTH | one year
  Show that patients receiving a dose of complete PTH 1-84 (CAP) and the ratio PTH 1-84/7-84 more easily reach the objectives international guidelines on the three following parameters calcium and phosphate: phosphorus, corrected calcium and phosphorus product.
  For each patient, a score will be awarded based on the number of criteria (including calcium, phosphorus and calcium phosphate product) in the target international guidelines:0-1-2 or 3.